CLINICAL TRIAL: NCT01418781
Title: Development of CLinical Prediction Rule Score in Veterans: A Study of Impact of Gout on Health Care Utilization and Costs
Brief Title: CLinical Prediction Rule Score in Veterans
Status: Withdrawn | Type: Observational
Why Stopped: Funding withdrawn by the funding agency; study could not be performed.
Sponsor: jasvinder singh (U.S. Federal Agency)
Collaborators: Birmingham, Alabama VA Medical Center (U.S. Federal Agency); Takeda (Industry); Novartis (Industry); Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, jasvinder singh, Worker without compensation, Minneapolis Veterans Affairs Medical Center
Organization: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Other Study IDs: MVAMC-3669A
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Gout
Keywords: gout; cost; utilization
MeSH Terms: conditions — Gout; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Gout: Patients with ICD-9 for gout
- No Gout: Patients withOUT ICD-9 for gout
- Tophaceous gout: Patients with ICD-9 for tophaceous gout
- non-tophaceous gout: those with ICD-9 for gout other than the codes specific for tophaceous gout

SUMMARY:
We will study whether the health care costs and health utilities differ in patients with gout and those without gout and whether they differ between those with more severe versus less severe gout

DETAILED DESCRIPTION:
The purpose of this project is to study the out-patient and inpatient utilization and costs associated with tophaceous gout (a classic form of treatment-failure gout), compare these costs to patients with non-tophaceous gout and evaluate health utilities associated with these gout states. The analyses will be conducted in a manner to support a burden of illness type of presentation / manuscript.

Study Questions

1. What are the VA health care costs (inpatient and outpatient) for patients with gout compared to those without gout?
2. Does health utility, as calculated by SF-6D, differ in patients with gout compared to patients without gout and between tophaceous and non-tophaceous gout?
3. What are the relationships between costs and health utility?
4. How does the burden of illness differ by subgroups of gout patients (costs and utilities)?
5. What are the VA health care costs for patients with tophaceous gout and are they higher than patients with non-tophaceous gout?

Inclusion criteria Patients with and without gout from the Veterans database described above will be included in the analyses for Study aims 1 and 5. This is approximately 3000 gout patients and 67,000 non-gout patients

Patients with SF-36 data from the above cohort will be included in the analyses for Study aims 2-4. This is approximately 1500 gout patients and 38,000 non-gout patients

ELIGIBILITY:
Inclusion Criteria:

* participated in the survey
* Have SF-36 adn utilization data

Exclusion Criteria:

* Absence of utilization and/or cost data

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with and without gout from the Veterans Upper Midwest SF-36 survey database will be included in the analyses for Study questions 1 and 5. This is approximately 3000 gout patients and 67,000 non-gout patients Patients with SF-36 data from the above cohort will be included in the analyses for Study aims 2-4. This is approximately 1500 gout patients and 38,000 non-gout patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Health care costs | Up to 5-year post-survey
  Total of outpatient, inpatient and emergent care costs

SECONDARY OUTCOMES:
Health utility index, SF-6D | 18-months
  at 18-month post-survey
Health care utilization | 1-year post-survey
  Health care utilization as sum of outpatient, inpatient and emergent care utilization
Activity limitation on Katz 6 ADL | 18-months
  Katz 6 ADL questions assess difficulty with doing 6 key activities, bathing, eating, toileting, walking, getting up and climbing stairs
Mortality | 5-years
  Up to 5-year post-survey

CONTACTS AND LOCATIONS:
Overall Officials: David Nelson, Principal Investigator — Minneapolis VAMC
Locations (1):
- Minneapolis VA Medical Center, Minneapolis, Minnesota, United States